CLINICAL TRIAL: NCT02445287
Title: Clinical Evaluation of CARESTREAM Cone Beam Computed Tomography (CBCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 6M3388
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Predicate & Invest.- Cadavers 2D & 3D (Experimental): Radiation - Cadaveric specimens will be imaged with 2D devices: CARESTREAM DRX-Evolution general radiograph and CARESTREAM Cone Beam Computed Tomography (CBCT) general radiograph, and 3D devices PHILLIPS Multi Detector Computed Tomography (MDCT) and CARESTREAM Cone Beam Computed Tomography (CBCT).
  Interventions: Radiation: Radiation
- Investigational - Human Subjects 3D (Experimental): Radiation - Human subjects will be imaged with 3D investigational device CARESTREAM Cone Beam Computed Tomography (CBCT) only.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Cadaveric specimens will be imaged with 2D devices: CARESTREAM DRX-Evolution general radiograph and CARESTREAM Cone Beam Computed Tomography (CBCT) general radiograph, and 3D devices PHILLIPS Multi Detector Computed Tomography (MDCT) and CARESTREAM Cone Beam Computed Tomography (CBCT). Human subjects will be imaged with CARESTREAM Cone Beam Computed Tomography (CBCT) 3D only.

SUMMARY:
The purpose of this study is to evaluate the 2D and 3D imaging performance of the CARESTREAM Cone Beam Computed Tomography (CBCT) scanner ("investigational device") against the commercially available 2D and 3D predicate devices. The results of this study will be included in a Traditional 510(k) FDA Submission to obtain clearance to market the new CARESTREAM Cone Beam Computed Tomography (CBCT) scanner in the US. The study was designed in accordance with the FDA Guidance titled "Guidance for the Submission of 510(k)'s for Solid State X-ray Imaging Devices", issued on August 6, 1999.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the 2D and 3D imaging performance of the CARESTREAM Cone Beam Computed Tomography (CBCT) scanner ("investigational device") against the commercially available 2D and 3D predicate devices. The study undertaken will demonstrate the safety and effectiveness of the investigational CARESTREAM Cone Beam Computed Tomography (CBCT) 2D imaging functionality by comparing against the predicate CARESTREAM DRX-1 GOS detector used on adult cadaver specimens to capture the image pairs.

The study will demonstrate the safety and effectiveness of the investigational CARESTREAM Cone Beam Computed Tomography (CBCT) 3D imaging functionality by comparing against the reference PHILLIPS Multi Detector Computed Tomography (MDCT) scanner used on adult cadaver specimens (body part) to capture 3D volumetric exams using the anatomy of both upper and lower extremity specimens. The adult cadaver specimens will receive multiple x-ray exposures using the predicate devices for both 2D and 3D imaging. Target images from cadaver specimens will be reviewed by radiologist readers to rate diagnostic image quality, and the data will be included in a comparative evaluation.

The live human subject portion of the study will be performed on healthy volunteers. Each volunteer will sign an Informed Consent after which will receive only one 3D volumetric exam using the investigational CARESTREAM Cone Beam Computed Tomography (CBCT) scanner. Target images will be reviewed by radiologist readers to rate diagnostic image quality according to a radiologist reader scale applicable to 3D volumetric imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years or older
* Subject has provided informed consent
* Subject is able to be positioned properly in the investigational device and be still during the exam to reduce the potential of motion in the images.
* Subject(s) may have a metal screw, plate or artificial joint

Exclusion Criteria:

* Subject is pregnant
* Not able or willing to provide Informed Consent, or consent is withdrawn
* Not able to collect all required case information
* Subject has a history of high radiation exposure:
* Has undergone radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Marzo, MD, Principal Investigator — UBMD Orthopaedics & Sports Medicine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Predicate & Invest.- Cadavers 2D & 3D: Cadaveric specimens will be imaged with 2D devices CARESTREAM DRX-Evolution general radiograph and CARESTREAM Cone Beam Computed Tomography (CBCT) general radiograph, and 3D devices PHILLIPS Multi Detector Computed Tomography (MDCT) and CARESTREAM Cone Beam Computed Tomography (CBCT).
- Investigational - Human Subjects 3D: Human subjects will be imaged with 3D investigational device CARESTREAM Cone Beam Computed Tomography (CBCT) only.
Period: Overall Study
Arm/Group | Predicate & Invest.- Cadavers 2D & 3D | Investigational - Human Subjects 3D
Started | 35 | 13
Completed | 35 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2D predicate and 3D reference devices were used on cadaveric specimens. Investigational CBCT 3D was used to image live humans.
Groups:
- Predicate & Invest.- Cadavers 2D & 3D: Cadaveric specimens will be imaged with 2D predicate device CARESTREAM DRX-1 GOS general radiograph and 2D investigational device CARESTREAM CBCT general radiograph. Cadaveric specimens will be imaged with 3D reference device Phillips MDCT and 3D investigational device CARESTREAM CBCT.
- Investigational - Human Subjects 3D: Human subjects will be imaged with 3D investigational device CARESTREAM CBCT only.
- Total: Total of all reporting groups
Arm/Group | Predicate & Invest.- Cadavers 2D & 3D | Investigational - Human Subjects 3D | Total
Number analyzed (Participants) | 35 | 13 | 48
Age, Customized [Number; unit: participants]
  18 years or older | 35 | 13 | 48
Sex/Gender, Customized [Number; unit: participants] — gender not collected for human subjects or cadaveric specimens
  participants
    Gender Unknown (not collected) | 35 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - 2D Images
Description: 1-1.9-Non-diagnostic Unacceptable for diagnostic purposes. Little or no clinically usable diagnostic information (e.g., gross underexposure, system failure or extensive motion artifact). Almost all such imaging should be repeated. 2-2.9-Limited Acceptable, with some technical defect (motion artifact, body habitus/poor x-ray penetration, or patient positioning may limit visualization of some body-regions but still adequate for diagnostic purposes). Not as much diagnostic information as is typical for an examination of this type, but likely sufficient. 3-3.9-Diagnostic Image quality that would be expected routinely when imaging cooperative patients. 4-Exemplary Good, most adequate for diagnostic purposes. Image quality that can serve as an example that should be emulated.
Time Frame: 12 weeks after last image capture
Population: 140 total image ratings from 4 radiologist readers (35 specimens rated x 4 readers) for each of the above two arms.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Groups:
- Predicate - Cadavers 2D; Investigational - Cadavers 2D: The study arms are broken out by participants which include cadaveric specimens imaged on both 2D (predicate and investigational) devices and 3D (reference and investigational) devices; and human subjects on 3D investigational device only. The image data is analyzed by comparing the following: 2D images from the predicate device to 2D images of the investigational device, and 3D images from the reference device to 3D images of the investigational device. In addition, the CBCT 3D device has three separate reconstructions that are available, high resolution iterative, Feldkamp, Davis & Kress (FDK), and standard iterative (SND). Therefore the outcome measures required four separate analyses (one for 2D and three for 3D) and are listed accordingly.
  All p-values were calculated (and verified) by our statistician and are correct. They were rounded to fit four digits.
Arm/Group | Predicate - Cadavers 2D | Investigational - Cadavers 2D
Number analyzed (Participants) | 35 | 35
Number analyzed (images) | 140 | 140
units on a scale | 3.4093 (0.0601) | 3.4179 (0.0602)
Statistical Analysis 1: Comparison: Predicate - Cadavers 2D vs Investigational - Cadavers 2D; Test type: Superiority or Other; p = 0.920, t-test, 2 sided — Level of significance (alpha) = 0.05

2. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - 3D Images High Resolution
Description: as for outcome 1
Time Frame: 12 weeks after last image capture
Population: 140 image ratings from 4 radiologist readers (35 specimens rated x 4 readers) for the for Reference-Cadavers 3D arm above. 204 image ratings from 4 radiologist readers (35 specimens, + 13 human subjects, + 3 specimens w/o metal correction rated x 4 readers) for the Investigational-Cadavers & Human Subjects 3D-High Resolution arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Groups:
- Reference - Cadavers 3D; Invest. - Cadavers & Human Subjects 3D - High Res: The study arms are broken out by participants which include cadaveric specimens imaged on both 2D (predicate and investigational) devices and 3D (reference and investigational) devices; and human subjects on 3D investigational device only. The image data is analyzed by comparing the following: 2D images from the predicate device to 2D images of the investigational device, and 3D images from the reference device to 3D images of the investigational device. In addition, the CBCT 3D device has three separate reconstructions that are available, high resolution iterative, Feldkamp, Davis & Kress (FDK), and standard iterative (SND). Therefore the outcome measures required four separate analyses (one for 2D and three for 3D) and are listed accordingly.
  All p-values were calculated (and verified) by our statistician and are correct. They were rounded to fit four digits.
Arm/Group | Reference - Cadavers 3D | Invest. - Cadavers & Human Subjects 3D - High Res
Number analyzed (Participants) | 35 | 48
Number analyzed (images) | 140 | 204
units on a scale | 3.5457 (0.0316) | 3.8377 (0.0211)
Statistical Analysis 1: Comparison: Reference - Cadavers 3D vs Invest. - Cadavers & Human Subjects 3D - High Res; Test type: Superiority or Other; p = 0.000, t-test, 1 sided — Level of significance (alpha) = 0.05

3. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - 3D Images FDK
Description: as for outcome 1
Time Frame: 12 weeks after last image capture
Population: 140 image ratings from 4 radiologist readers (35 specimens rated x 4 readers) for the for Reference-Cadavers 3D arm above. 204 image ratings from 4 radiologist readers (35 specimens, + 13 human subjects, + 3 specimens w/o metal correction rated x 4 readers) for the Investigational-Cadavers & Human Subjects 3D-FDK arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Groups:
- Invest. - Cadavers & Human Subjects 3D - FDK: The study arms are broken out by participants which include cadaveric specimens imaged on both 2D (predicate and investigational) devices and 3D (reference and investigational) devices; and human subjects on 3D investigational device only. The image data is analyzed by comparing the following: 2D images from the predicate device to 2D images of the investigational device, and 3D images from the reference device to 3D images of the investigational device. In addition, the CBCT 3D device has three separate reconstructions that are available, high resolution iterative, Feldkamp, Davis & Kress (FDK), and standard iterative (SND). Therefore the outcome measures required four separate analyses (one for 2D and three for 3D) and are listed accordingly.
  All p-values were calculated (and verified) by our statistician and are correct. They were rounded to fit four digits.
Arm/Group | Reference - Cadavers 3D | Invest. - Cadavers & Human Subjects 3D - FDK
Number analyzed (Participants) | 35 | 48
Number analyzed (images) | 140 | 204
units on a scale | 3.5277 (0.0316) | 3.5353 (0.0372)
Statistical Analysis 1: Comparison: Reference - Cadavers 3D vs Invest. - Cadavers & Human Subjects 3D - FDK; Test type: Non-Inferiority or Equivalence — Equivalence interval = (-0.25, 0.25); p = 0.000, Equivalence test — level of significance (alpha) = 0.05

4. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - 3D Images SND
Description: as for outcome 1
Time Frame: 12 weeks after last image capture
Population: 140 image ratings from 4 radiologist readers (35 specimens rated x 4 readers) for the for Reference-Cadavers 3D arm above. 204 image ratings from 4 radiologist readers (35 specimens, + 13 human subjects, + 3 specimens w/o metal correction rated x 4 readers) for the Investigational-Cadavers & Human Subjects 3D-SND arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Groups:
- Invest. - Cadavers & Human Subjects 3D - SND: The study arms are broken out by participants which include cadaveric specimens imaged on both 2D (predicate and investigational) devices and 3D (reference and investigational) devices; and human subjects on 3D investigational device only. The image data is analyzed by comparing the following: 2D images from the predicate device to 2D images of the investigational device, and 3D images from the reference device to 3D images of the investigational device. In addition, the CBCT 3D device has three separate reconstructions that are available, high resolution iterative, Feldkamp, Davis & Kress (FDK), and standard iterative (SND). Therefore the outcome measures required four separate analyses (one for 2D and three for 3D) and are listed accordingly.
  All p-values were calculated (and verified) by our statistician and are correct. They were rounded to fit four digits.
Arm/Group | Reference - Cadavers 3D | Invest. - Cadavers & Human Subjects 3D - SND
Number analyzed (Participants) | 35 | 48
Number analyzed (images) | 140 | 204
units on a scale | 3.5277 (0.0316) | 3.6319 (0.0333)
Statistical Analysis 1: Comparison: Reference - Cadavers 3D vs Invest. - Cadavers & Human Subjects 3D - SND; Test type: Superiority or Other; p = 0.012, t-test, 1 sided — level of significance (alpha) = 0.05

ADVERSE EVENTS:
Time Frame: AE's were collected for 3 months, September - November 2015
Groups:
- Predicate & Invest.- Cadavers 2D: Cadaveric specimens will be imaged with 2D predicate device CARESTREAM DRX-1 GOS general radiograph and 2D investigational device CARESTREAM CBCT general radiograph.
- Reference & Invest. - Cadavers 3D: Cadaveric specimens will be imaged with 3D reference device Phillips MDCT and 3D investigational device CARESTREAM CBCT.
Arm/Group | Predicate & Invest.- Cadavers 2D | Reference & Invest. - Cadavers 3D | Investigational - Human Subjects 3D
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/13
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No